CLINICAL TRIAL: NCT02183207
Title: Percutaneous Endoscopic Gastrostomy by Introducer Method Via Visualization Through E.G. ScanTM
Brief Title: PEG by Introducer Method Via EG Scan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Collaborators: IntroMedic Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Myung-gui Choi, Professor, The Catholic University of Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEG by EG Scan
Record Dates: First submitted 2013-08-11; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Dysphagia; Aspiration; Esophageal Stenosis
Keywords: percutaneous endoscopic gastrostomy; Introducer method
MeSH Terms: conditions — Deglutition Disorders; Esophageal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PEG insertion arm via EG Scan (Experimental): Percutaneous endoscopic insertion of gastrostomy via visualization through E.G. ScanTM
  Interventions: Procedure: Percutaneous Endoscopic Gastrostomy

INTERVENTIONS:
Procedure: Percutaneous Endoscopic Gastrostomy — Percutaneous Endoscopic Gastrostomy by introducer method via visualization through E.G. ScanTM

SUMMARY:
Percutaneous endoscopic gastrostomy(PEG) by introducer method has been proven to be safe and easy to perform. However, it is limited by its need to be performed in an endoscopy unit. E.G. ScanTM is an new portable ultrathin endoscope, capable of being performed in any hospital setting and introduced via nasal approach. Our aim is to prove that PEG by introducer method via E.G. ScanTM is feasible and safe. This will allow PEG to be done at hospitals and medical facilities without endoscopic units.

ELIGIBILITY:
Inclusion Criteria:

* Require percutaneous endoscopic gastrostomy placement due to inability to achieve oral feeding for at least one month

Exclusion Criteria:

* Patients with esophageal ulcers or strictures
* Patients with prior esophageal/gastric surgery (excepting gastric wedge resection)
* Patients at high risk of gastric bleeding, mechanical ileus or gastrointestinal perforation
* Other patients in whom the study investigators consider unfit for inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-07 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
The success rate of PEG via introducer method by visualization through EG ScanTM | up to 1 year from PEG insertion
  up to 1 year from PEG insertion or until patient death if within one year

SECONDARY OUTCOMES:
Complication rate | up to one year from PEG insertion
  Complication rate including bleeding, infection, gastric perforation and leakage of intragastric contents

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul St Mary's Hospital, Seoul, South Korea

REFERENCES:
- [Result] Dormann AJ, Wejda B, Kahl S, Huchzermeyer H, Ebert MP, Malfertheiner P. Long-term results with a new introducer method with gastropexy for percutaneous endoscopic gastrostomy. Am J Gastroenterol. 2006 Jun;101(6):1229-34. doi: 10.1111/j.1572-0241.2006.00541.x. PMID 16771943
- [Result] Yuki M, Amano Y, Komazawa Y, Fukuhara H, Shizuku T, Yamamoto S, Kinoshita Y. Unsedated transnasal small-caliber esophagogastroduodenoscopy in elderly and bedridden patients. World J Gastroenterol. 2009 Nov 28;15(44):5586-91. doi: 10.3748/wjg.15.5586. PMID 19938199